CLINICAL TRIAL: NCT00975858
Title: A Randomized Comparison of Long-term Clinical , Neurocognitive, Angiographical and Health-costs, After Stenting Versus Off-pump Coronary Bypass Surgery in Patients With Symptomatic Coronary Artery Disease
Brief Title: Long-term Comparison of Stenting Versus Off-pump Coronary Bypass Surgery
Acronym: OCTOSTENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: St. Antonius Hospital (Other); Isala (Other)
Responsible Party: JJ Regiel, MD / HM Nathoe, MD,PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WOM protocol 98/009
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Artery Disease
Keywords: Symptomatic Coronary Artery Disease Patients
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous Coronary Intervention (Active Comparator)
  Interventions: Procedure: Coronary Revascularization
- Off Pump Coronary Artery Bypass Surgery (Experimental)
  Interventions: Procedure: Coronary Revascularization

INTERVENTIONS:
Procedure: Coronary Revascularization — revascularization of coronary arteries in case of symptomatic obstructive coronary artery disease
  Other Names: Stenting; PCI; OPCAB; MICAB

SUMMARY:
The randomized comparison of two strategies in coronary revascularization: bypass surgery without the use of a heart lung machine and coronary stenting procedure.

The comparison comprised the occurrence of cardiac adverse events after the procedure. In addition, costs, cognitive outcomes and angiography were assessed.

DETAILED DESCRIPTION:
Coronary artery bypass surgery with use of the heart lung machine (on-pump surgery), is associated with the risk of peri-operative complications such as death, stroke, myocardial infarction, neurocognitive decline, and extended hospitalization. Bypass surgery on the beating heart without the use of the heart lung machine (off-pump surgery) has been reintroduced in clinical practice in order to reduce these complications. The Octopus cardiac wall stabilizer, developed at the UMC Utrecht, facilitates the safe construction of the grafts during the off-pump procedure. The expected advantages of off-pump surgery e.g. less-invasiveness, complete arterial revascularization, faster recovery and lower costs were the basis for the Octostent trial. We hypothesized that the off-pump surgical technique might offer an alternative for angioplasty with bare-metal stent-implantation.

The current study was designed as a randomized controlled multicenter trial comparing two strategies.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease referred for PCI in which both Off Pump Coronary Bypass surgery and PCI were deemed technically feasible

Exclusion Criteria:

* a history of CABG or stenting
* emergency or concomitant major surgery
* Q-wave myocardial infarction in the last six weeks
* inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 1998-01; Primary Completion 2001-01 (Actual); Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 7.5 years

SECONDARY OUTCOMES:
Quality of Life | 7.5 years
Neurocognitive outcome | 7.5 years
Cost effectiveness | 7.5 years
Angiographical patency of revascularization | 7.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik M Nathoe, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Eefting F, Nathoe H, van Dijk D, Jansen E, Lahpor J, Stella P, Suyker W, Diephuis J, Suryapranata H, Ernst S, Borst C, Buskens E, Grobbee D, de Jaegere P. Randomized comparison between stenting and off-pump bypass surgery in patients referred for angioplasty. Circulation. 2003 Dec 9;108(23):2870-6. doi: 10.1161/01.CIR.0000100723.50363.2C. Epub 2003 Dec 1. PMID 14656913